CLINICAL TRIAL: NCT06187623
Title: COMPARISON OF THE EFFECTIVENESS OF CLINICAL AND HOME-BASED SCHROTH EXERCISES ON ADOLESCENT IDIOPATHIC SCOLIOSIS INDIVIDUALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Ipek Yurttaş, Physiotherapist, Uskudar University
Other Study IDs: Physiotherapy rehabilitation
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: scoliosis; brace; exercise; proprioception; neck
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Home based Group: 15 patients in the home-based group and their parents will be informed about the treatment program. Exercise training will be given to individuals by a physiotherapist trained in ISST- International Schroth 3-Dimensional Scoliosis Therapy.
  Individuals in this group will be included in an exercise program 1 day a week (8 sessions) accompanied by a physiotherapist for 8 weeks. Each exercise session will last 50 minutes. Patients will be asked to do the given home exercises on the remaining 6 days of the week.
  Interventions: Other: Home based exercise
- Clinic based Group: 15 patients and their parents in the clinic-based group will be informed about the treatment program. Exercise training will be given to individuals by a physiotherapist trained in ISST- International Schroth 3-Dimensional Scoliosis Therapy.
  Individuals in this group will be included in an exercise program 3 days a week (24 sessions) with a physiotherapist for 8 weeks. Each exercise session will last 50 minutes. Patients will be asked to do the given home exercises on the remaining 4 days of the week.
  Interventions: Other: Clinic based exercise

INTERVENTIONS:
Other: Clinic based exercise — 15 patients and their parents in the clinic-based group will be informed about the treatment program. Exercise training will be given to individuals by a physiotherapist trained in ISST- International Schroth 3-Dimensional Scoliosis Therapy.
  Individuals in this group will be included in an exercise program 3 days a week (24 sessions) with a physiotherapist for 8 weeks. Each exercise session will last 50 minutes. Patients will be asked to do the given home exercises on the remaining 4 days of the week.
  Groups: Clinic based Group
Other: Home based exercise — 15 patients in the home-based group and their parents will be informed about the treatment program. Exercise training will be given to individuals by a physiotherapist trained in ISST- International Schroth 3-Dimensional Scoliosis Therapy.
  Individuals in this group will be included in an exercise program 1 day a week (8 sessions) accompanied by a physiotherapist for 8 weeks. Each exercise session will last 50 minutes. Patients will be asked to do the given home exercises on the remaining 6 days of the week.
  Groups: Home based Group

SUMMARY:
In individuals diagnosed with AIS, significant regressions in curvature were observed with the use of schroth exercises and brace. It is known that neurological changes affect the vestibular system and create changes in the individual's balance and proprioception. At the same time, when static and balance are examined, it is seen that they have difficulty in maintaining their dynamic balance and their body center of gravity oscillations increase. There are a limited number of studies in the literature evaluating individuals diagnosed with AIS in the combined treatment of brace use and Schroth exercises.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of clinic and home-based Schroth exercises in individuals diagnosed with adolescent idiopathic scoliosis.

The 30 participants who will participate in the study will be between the ages of 10-18 and their Cobb angle will vary between 25-45 degrees. Consent forms will be obtained from all participants participating in the study.

Cervical Relocation Test to measure participants' proprioception; Y-Balance Test will be used for dynamic balance, evaluation of trunk rotation angle with a scoliometer, Spinal Appearence Questionnaire for cosmetic deformity perception, Bad-Sobernheim Stress Questionnaire will be used for brace stress.

Demographic information such as age (years), weight (kg), height (cm), lower extremity length (cm), primary curvatures, daily brace use time (hours), brace use frequency of the people who agreed to participate in the study were collected. corset revision The number and use of insoles (yes or not) will be questioned.

The Cervicocephalic Relocation Test developed by Revel will be used to evaluate cervical proprioception. Blindfolded subjects will be seated on a chair with a backrest, 90cm away from the wall on which a circular target board is hung. They will be asked to sit as far back in the chair as possible, placing their arms on their laps, and leaning on the back of the chair. Each subject has a laser pointer attached to their head and their eyes will be covered with a sleep mask. The person's head position will be placed on the target board by the therapist, showing the laser zero point, and 5 seconds will be given to remember this point. Subjects will experience the test with their eyes open before starting the experiment. After concentrating on this reference position for a few seconds, the patient will be asked to move the head in the previously shown directions (flexion, extension) for 5 repetitions and return to the reference point. The distance between the starting head position and the ending head position will be calculated as the angular result by placing it in the formula angle = tan -1 [Distance between the start and the end cm/90 cm].

Dynamic Balance- Y Balance Test After the foot of the party to be tested is placed behind the red line on the platform, they will be asked to push the distance indicator in all three directions (anterior, postromedial and posterolateral) as far as possible with the foot in the air. After two trials are made in each direction before the test, three measurements will be taken for each direction during the test phase. For each direction, the total score obtained by dividing the best value of the three maximum distances by the leg length and multiplying by 100 will be calculated and noted. The test will be terminated when the person lifts the heel of the tested foot standing on the platform to maintain balance during the test, loses contact with the distance indicator, uses it as support to restore the lost balance and cannot return to the starting position.

Scoliometer, individuals will be asked to stand upright, looking forward with their feet parallel and adjacent to each other, and then the individual will be told that they should lean forward with their hands and feet together, keeping their body parallel to the ground. During the evaluation, the spinous processes will be monitored with a scoliometer, starting from the cervical region to the lumbar region.

For quality of life assessment; Bad Sobernheim Stress Questionnaire and Scoliosis Appearance Questionnaire were used. Evaluations will be answered twice, before and after.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 10-18,
* Being diagnosed with Adolescent Idiopathic Scoliosis (AIS),
* COBB angles should be between 20 and 45 degrees,
* Risser sign being between 0-5,
* Having brace treatment given by the doctor.

Exclusion Criteria:

* Having a different diagnosis such as congenital scoliosis, spina bifida, traumatic scoliosis, osteoporosis,
* Having had spine surgery,
* Stating that you will not comply with the corset period prescribed by the doctor,
* Having serious cardiopulmonary problems that will prevent them from exercising,
* Individuals and parents did not agree to sign the consent form required to participate in the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: ınviduals between the ages of 10-18 who have been diagnosed with AIS and having brace treatment given by the doctor come to our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-03-04 (Estimated)

PRIMARY OUTCOMES:
The effect of clinical based Schroth exercises on the cervical proprioception | 15 minutes
  Individuals will be seated with their eyes closed, with the laser pointer on their heads, and will be asked to target the 0 point on the target board in front of them. After performing 5 repetitions of flexion and 5 repetitions of extension movements, deviations from the 0 point will be recorded.
The effect of home based Schroth exercises on the cervical proprioception | 15 minutes
  Individuals will be seated with their eyes closed, with the laser pointer on their heads, and will be asked to target the 0 point on the target board in front of them. After performing 5 repetitions of flexion and 5 repetitions of extension movements, deviations from the 0 point will be recorded.

SECONDARY OUTCOMES:
The effect of home based Schroth exercises on the dynamic balance | 10 minutes
  The lower extremity to be evaluated is lifted onto the testing platform. It is desired to extend to the anterior, posterolateral and posteromedial directions, respectively. The longest distance it can reach is recorded.
The effect of clinic based Schroth exercises on the dynamic balance | 10 minutes
  The lower extremity to be evaluated is lifted onto the testing platform. It is desired to extend to the anterior, posterolateral and posteromedial directions, respectively. The longest distance it can reach is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ipek yurttaş, Principal Investigator — Üsküdar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No